CLINICAL TRIAL: NCT04664751
Title: Incidence of Compliance to the ASA Preoperative Fasting Guidelines in Elective General Surgery.
Brief Title: Incidence of Compliance to the ASA Preoperative Fasting Guidelines in Elective Surgery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Other Study IDs: 997/2563(IRB2)
Record Dates: First submitted 2020-11-25; First posted 2020-12-11 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Compliance, Treatment
Keywords: Compliance; NPO guidelines
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients scheduled for general surgery with anesthesia: Patients scheduled for general surgery with anesthesia, receiving Nil-per-Oral order.
  Interventions: Other: Nil-per-Oral

INTERVENTIONS:
Other: Nil-per-Oral — NPO details

SUMMARY:
Patients scheduled for elective surgery with general anesthesia, regional anesthesia, or procedural sedation and analgesia will be interviewed about the last time having

* clear liquid drink
* light meal
* regular meal

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery requiring general anesthesia, regional anesthesia, or procedural sedation and analgesia.

Exclusion Criteria:

* Patients with the order of NPO after midnight.
* Patients with pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery requiring general anesthesia, regional anesthesia, or procedural sedation and analgesia
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
compliance to NPO guideline | 8 hour
  definition of compliance include complete order of NPO for regular diet for 8 hours and soft diet for 6 hours and clear liquid for 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No